CLINICAL TRIAL: NCT06476938
Title: Testing the Efficacy of an eHealth Decision Support Tool to Help Latinx Cancer Patients Make Informed Decisions About Tumor Genomic Testing
Brief Title: Testing Gene PilotLX With Latinx Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Temple University (Other); MD Anderson Cancer Center at Cooper (Other); Herbert Irving Comprehensive Cancer Center (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-1047; U54CA221705 (NIH)
Record Dates: First submitted 2024-06-17; First posted 2024-06-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Cancer
Keywords: eHealth decision tool; Hispanic/Latino; Tumor Genomic Profiling
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gene PilotLX (Experimental): Gene PilotLX is an eHealth decision support tool that is designed to empower Latinx cancer patients to decide their preferences for learning about secondary genetic information, communicate those preferences to their doctors, and provide the opportunity to discuss information with their families or others to feel they have made an informed decision. The tool will be available in both English and Spanish. It is web-based, has a voice-over, and is easy to navigate, with simple forward and backward buttons. Each section includes a different aspect of tumor genomic profiling, from basic information about what the test is and what the pros and cons are of the test, to culturally specific potential barriers or benefits to learning hereditary results. At the end, the tool provides tailored potential questions for a doctor that users can choose, which are summarized in a "score card" that can be printed or emailed.
  Interventions: Other: Gene PilotLX
- TGP brochure (No Intervention): Participants in the control arm will be provided a brochure about tumor genomic profiling (TGP) secondary hereditary risks, and what patients can decide about getting that information, including the pros and cons. It is literacy appropriate, incorporates visuals, and will also be offered in both English and Spanish.

INTERVENTIONS:
Other: Gene PilotLX — eHealth decision making tool regarding tumor genomic profiling
  Arms: Gene PilotLX

SUMMARY:
This is a randomized controlled trial designed to evaluate the efficacy of an electronic health decision support tool called Gene PilotLX to increase informed decision making regarding hereditary risk information from tumor genomic profiling (TGP) test among Latinx cancer patients recruited at four cancer centers.

DETAILED DESCRIPTION:
The use of multi-gene tumor genomic profiling (TGP) to examine a patient's tumor for targetable mutations is a cornerstone of personalized oncology. Providers are required to communicate TGP risks to patients and elicit patient preferences for managing information (i.e., "opt out" or have genetic counseling) because of the possibility of uncovering secondary hereditary cancer risks found on this test. Yet barriers exist to support optimal decision-making. Limited study of genetic links to cancer has been done with Latinx patients making them an important understudied group to target for genetic decision support. Shared cultural values among Latinx individuals such as familismo (family loyalty) and fatalismo (fatedness) may influence how patients approach cancer risk assessment and genetics and language and acculturation barriers, access and affordability, deportation risks, medical mistrust and low genetic knowledge impact decision making. As a result, Latinx patients are less likely to participate in clinical genetic testing. Adding to this vulnerability is the fact that many oncologists may not have a good understanding of how to effectively communicate secondary hereditary risks to Latinx patients. This leaves Latinx patients without the support they need to make good decisions about what they would want to do about secondary results from TGP that is in line with their needs, preferences and values.

eHealth interventions can promote health behavior change when developed with targeted messages, but many fall short if they do not effectively address the core barriers to a health decision. Gene PilotLX was developed using commercial marketing techniques to ensure saliency. Using perceptual mapping and vector message modeling, the investigators have shown in our parent Gene Pilot study that was conducted among AA/Black cancer patients that this approach provides a superior methodology for developing effective, persuasive messages that result in significant behavior and decisional conflict changes.

A fully powered randomized controlled trial will be conducted with 232 Latinx cancer patients at four oncology sites to evaluate the efficacy of Gene PilotLX,an electronic health decision support tool. Participants will be randomized either to intervention arm and watch Gene PilotLX or usual arm and review patient information about TGP presented in a written document (pdf). All participants will complete three assessments: baseline, immediate post intervention, and 1-3-month surveys.

ELIGIBILITY:
Inclusion Criteria:

Self-identified Latinx patients who:

1. diagnosed with solid tumor cancers
2. speak/read English or Spanish;
3. can provide informed consent.

Exclusion Criteria:

Patients with hematologic/liquid cancers (leukemia, lymphoma, multiple myeloma, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Preparation for Decision Making (PrepDM) Scale | Post-test (can occur on same day as baseline, day 1) and 1-3 month follow-up
  PrepDM Scale measures preparedness of patient to make a decision (10 items) regarding a hereditary risk from tumor genomic profiling (TGP) on a 1 "not at all" to 5 "a great deal" scale. Higher means indicated higher perceived level of preparation for decision making.
Decisional Conflict: Ottawa Decision Support Framework (ODSF) scale | Post-test (can occur on same day as baseline, day 1) and 1-3 month follow-up
  16- item measure to determine patient clarity on the risks and benefits of tumor genomic profiling (TGP) testing and hereditary risk information from TGP. Items are given a score value of: 0= 'strongly agree'; 2= 'neither agree nor disagree'; 3= 'disagree'; 4= 'strongly disagree' TOTAL SCORE 16 items are: a) summed; b) divided by 16; and c) multiplied by 25. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict]
Communication of preferences to doctor related to pursuing hereditary cancer risk information from TGP | 1-3 month follow up
  This is a single dichotomous item created for the study: 'Have you talked with a doctor about secondary hereditary results from TGP testing'?('Yes', 'No'). If 'Yes' is selected, 7 different topics for discussion with doctor are listed, including 'other' as open question.

SECONDARY OUTCOMES:
Communication of preferences with family related to pursuing hereditary cancer risk information from TGP | 1-3 month follow up
  This is a single dichotomous item created for the study: 'Have you talked about secondary hereditary results from TGP testing with your family, friends or spouse/partner'? ('Yes', 'No'). If 'Yes' is selected, 7 different topics for discussion with family are listed, including 'other' as open question.
Perception of Tumor Genomic Profiling (TGP) | Baseline (day1) and 1-3 month follow up
  18 statements related to benefits and concerns of TGP were developed as part of formative work (focus group with patients) for our previous work with AA/Black cancer patients and are related to beliefs, perceived barriers and benefits of TGP testing; 0-10 agreement scale when 0 is 'strongly disagree' and 10 'strongly agree'. Perceptual maps will be generated from the survey responses. Perceptual mapping methods developed by co-PI Bass use multidimensional scaling (MDS) analysis to create 3-Dimensional representations of how participants conceptualizes a decision and then message vector modeling techniques are used to design messages that will be most likely to persuade participants to make that decision. This method will be used to design messages for Gene PilotLX, the eHealth decision aid for Latinx cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hall, MD,MS, Principal Investigator — Fox Chase Cancer Center; Sarah B Bass, PhD, MPH, Principal Investigator — Temple University; Tracey A Revenson, PhD, Principal Investigator — Hunter College of City University of New York
Locations (4):
- United States (4):
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catenacci DV, Amico AL, Nielsen SM, Geynisman DM, Rambo B, Carey GB, Gulden C, Fackenthal J, Marsh RD, Kindler HL, Olopade OI. Tumor genome analysis includes germline genome: are we ready for surprises? Int J Cancer. 2015 Apr 1;136(7):1559-67. doi: 10.1002/ijc.29128. Epub 2014 Aug 14. PMID 25123297
- [Background] Schrader KA, Cheng DT, Joseph V, Prasad M, Walsh M, Zehir A, Ni A, Thomas T, Benayed R, Ashraf A, Lincoln A, Arcila M, Stadler Z, Solit D, Hyman DM, Zhang L, Klimstra D, Ladanyi M, Offit K, Berger M, Robson M. Germline Variants in Targeted Tumor Sequencing Using Matched Normal DNA. JAMA Oncol. 2016 Jan;2(1):104-11. doi: 10.1001/jamaoncol.2015.5208. Erratum In: JAMA Oncol. 2016 Feb;2(2):279. doi: 10.1001/jamaoncol.2015.6541.. Hyman, David [corrected to Hyman, David M]. PMID 26556299
- [Background] Cruz-Correa M, Perez-Mayoral J, Dutil J, Echenique M, Mosquera R, Rivera-Roman K, Umpierre S, Rodriguez-Quilichini S, Gonzalez-Pons M, Olivera MI, Pardo S; Puerto Rico Clinical Cancer Genetics Consortia. Clinical Cancer Genetics Disparities among Latinos. J Genet Couns. 2017 Jun;26(3):379-386. doi: 10.1007/s10897-016-0051-x. Epub 2016 Dec 12. PMID 27957667
- [Background] Lynce F, Graves KD, Jandorf L, Ricker C, Castro E, Moreno L, Augusto B, Fejerman L, Vadaparampil ST. Genomic Disparities in Breast Cancer Among Latinas. Cancer Control. 2016 Oct;23(4):359-372. doi: 10.1177/107327481602300407. PMID 27842325
- [Background] Pagan JA, Su D, Li L, Armstrong K, Asch DA. Racial and ethnic disparities in awareness of genetic testing for cancer risk. Am J Prev Med. 2009 Dec;37(6):524-30. doi: 10.1016/j.amepre.2009.07.021. PMID 19944919
- [Background] Canedo JR, Miller ST, Myers HF, Sanderson M. Racial and ethnic differences in knowledge and attitudes about genetic testing in the US: Systematic review. J Genet Couns. 2019 Jun;28(3):587-601. doi: 10.1002/jgc4.1078. Epub 2019 Jan 21. PMID 30663831
- [Background] Furness K, Sarkies MN, Huggins CE, Croagh D, Haines TP. Impact of the Method of Delivering Electronic Health Behavior Change Interventions in Survivors of Cancer on Engagement, Health Behaviors, and Health Outcomes: Systematic Review and Meta-Analysis. J Med Internet Res. 2020 Jun 23;22(6):e16112. doi: 10.2196/16112. PMID 32574147
- [Background] Wagner LI, Tooze JA, Hall DL, Levine BJ, Beaumont J, Duffecy J, Victorson D, Gradishar W, Leach J, Saphner T, Sturtz K, Smith ML, Penedo F, Mohr DC, Cella D. Targeted eHealth Intervention to Reduce Breast Cancer Survivors' Fear of Recurrence: Results From the FoRtitude Randomized Trial. J Natl Cancer Inst. 2021 Nov 2;113(11):1495-1505. doi: 10.1093/jnci/djab100. PMID 34057469
- [Background] Wilson J, Heinsch M, Betts D, Booth D, Kay-Lambkin F. Barriers and facilitators to the use of e-health by older adults: a scoping review. BMC Public Health. 2021 Aug 17;21(1):1556. doi: 10.1186/s12889-021-11623-w. PMID 34399716